CLINICAL TRIAL: NCT04455412
Title: Laser Assisted ICSI; Has it Role Whatsoever? Does it Affect the ICSI Outcome Positively?1
Brief Title: Laser Assisted ICSI; Has it Role Whatsoever?
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment is stopped waiting for funds
Sponsor: Royal Fertility Center, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RoyalFertility 001
Record Dates: First submitted 2020-06-28; First posted 2020-07-02 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Laser Assistance to Improve ICSI Outcome
Keywords: Laser assisted-ICSI; Zona pellucida thinning; ICSI; embryo good quality rate; hatching rate

STUDY DESIGN:
Intervention Model Description: study divided into three interventions; Conventional ICSI (control group) was compared with LAD-ICSI (Study group 1) and LAT- ICSI (study group 2) in sibling oocytes. then Cases randomly selected for embryo transfer from each group
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- control group (No Intervention): Conventional ICSI procedure was done for first portion of sibling oocytes
- Study group 1 (Experimental): Laser assisted drilling ICSI procedure was done for second portion of sibling oocytes
  Interventions: Procedure: Laser Assisted ICSI
- Study group 2 (Experimental): Laser assisted thinning ICSI procedure was done for Third portion of sibling oocytes
  Interventions: Procedure: Laser Assisted ICSI

INTERVENTIONS:
Procedure: Laser Assisted ICSI — using OCTICS laser device to do small opening or zona thinning to improve ICSI outcome
  Arms: Study group 1; Study group 2

SUMMARY:
laser-assisted ICSI (LA-ICSI) was described to be a new method combining a less invasive ICSI technique with assisted hatching.This procedure is usually used for MII oocytes possessing oolemma breakage difficulties, but why not using it for even normal Oocytes?!. Especially because data indicated that in addition to an improved oocyte survival, this new approach increases the hatching rate in vitro. But since it is still debatable that such a small opening might impair the hatching process, so modified zona thinning technique was proposed for more embryo safety.

DETAILED DESCRIPTION:
This study aims to compare the LA- ICSI by drilling a micro hole (LAD-ICSI) and modified LA-ICSI by zona pellucida thinning (LAT-ICSI) with conventional ICSI in order to effectively assess whether this approach can be applied routinely to improve ICSI outcome.

One arm study divided into three interventions; Conventional ICSI (control group) was compared with LAD-ICSI (Study group 1) and LAT- ICSI (study group 2) in sibling oocytes.

The rates of maturation, fertilization, Devision, Blastulation and good quality blastulation rates were assessed in the three groups

Cases were randomly selected for embryo transfer from the three groups,Then chemical pregnancy and clinical pregnancy rates were compared between the three groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 20 years old to 37 years old
* good res-ponders
* gives more than 15 oocytes
* endometrial thickness more than 9 mm

Exclusion Criteria:

* poor res-ponders
* severe oligoasthinozoospermia of male partners
* testicular samples
* Poor quality oocytes

Ages: 20 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | three-four weeks after embryo transfer
  confirmed by sac observation using ultrasound

SECONDARY OUTCOMES:
Blastulation rate | 5 days later after ICSI procedure
  number of blastocysts that are grown from devided embryos
Hatching rate | 5 days later after ICSI procedure
  number of blastocysts that hatch out of zona

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Fertility Center, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No